CLINICAL TRIAL: NCT00617929
Title: Conditioning for Graft Failure After Hematopoietic Stem Cell Transplantation
Brief Title: Antithymocyte Globulin, Clofarabine, and Rituximab in Treating Patients After an Unsuccessful Stem Cell Transplant
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Replaced by another protocol
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007LS072; UMN-MT2007-07 (Other: Blood and Marrow Transplantation Program); 0707M11845 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2008-02-15; First posted 2008-02-18 (Estimated); Results first posted 2017-01-20 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Cancer
Keywords: chronic myelogenous leukemia; acute lymphoblastic leukemia; chronic myeloid leukemia; lymphoblastic leukemia; acute myeloid leukemia; chronic eosinophilic leukemia; primary myelofibrosis; chronic myelomonocytic leukemia; chronic neutrophilic leukemia; de novo myelodysplastic syndromes; disseminated neuroblastoma; juvenile myelomonocytic leukemia; Burkitt lymphoma; rhabdomyosarcoma; myelodysplastic syndromes; Hodgkin lymphoma; lymphoblastic lymphoma; breast cancer; follicular lymphoma; mantle cell lymphoma; marginal zone lymphoma; recurrent neuroblastoma; recurrent ovarian epithelial cancer; recurrent ovarian germ cell tumor; recurrent small lymphocytic lymphoma; recurrent malignant testicular germ cell tumor; recurrent Wilms tumor and other childhood kidney tumors; recurrent/refractory childhood Hodgkin lymphoma; refractory hairy cell leukemia; refractory multiple myeloma; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; splenic marginal zone lymphoma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; stage II ovarian epithelial cancer; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult Hodgkin lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III chronic lymphocytic leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III ovarian epithelial cancer; stage III small lymphocytic lymphoma; stage III malignant testicular germ cell tumor; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV breast cancer; stage IV chronic lymphocytic leukemia; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV ovarian epithelial cancer; stage IV small lymphocytic lymphoma; refractory chronic lymphocytic leukemia
MeSH Terms: conditions — Neoplasms; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic; Leukemia, Myelomonocytic, Juvenile; Burkitt Lymphoma; Rhabdomyosarcoma; Myelodysplastic Syndromes; Hodgkin Disease; Breast Neoplasms; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Neuroblastoma; Carcinoma, Ovarian Epithelial; Leukemia, Lymphocytic, Chronic, B-Cell; Testicular Neoplasms; Wilms Tumor; Recurrence; Leukemia, Hairy Cell; Multiple Myeloma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic | interventions — Antilymphocyte Serum; thymoglobulin; Rituximab; Clofarabine; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Conditioning for Graft Failure (Experimental): Primary or secondary graft failure after hematopoietic stem cell transplantation defined as a > 50% loss of previously best donor chimerism or less than 25% donor chimerism beyond day +42 with pancytopenia and no evidence of relapse. Patients with any diagnosis, type of donor, hematopoietic cell graft or conditioning regimen should be considered for this study. Patients receive anti-thymocyte globulin, rituximab, and clofarabine.
  Interventions: Biological: anti-thymocyte globulin; Biological: rituximab; Drug: clofarabine; Procedure: stem cell transplantation

INTERVENTIONS:
Biological: anti-thymocyte globulin — administer 3 mg/kg intravenously (IV) over 4 hours on days -6, -5 and -4.
  Other Names: Thymoglobulin®
Biological: rituximab — administered 375 mg/m^2 intravenously (IV) in 1 mg/mL normal saline on day -7.
  Other Names: Rituxan(R)
Drug: clofarabine — administered 30 mg/m^2 intravenously (IV) over 1 hour on Days -4, -3, and -2.
  Other Names: CLOLAR™
Procedure: stem cell transplantation — administered on Day 0 per institutional guidelines.

SUMMARY:
RATIONALE: Antithymocyte globulin, clofarabine, and rituximab may stop the patient's immune system from rejecting the donor's stem cells when they do not exactly match the patient's blood. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving antithymocyte globulin before transplant and cyclosporine and mycophenolate mofetil before and after transplant may stop this from happening.

PURPOSE: This phase II trial is studying how well giving antithymocyte globulin together with clofarabine and rituximab works in treating patients after an unsuccessful stem cell transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the rate of sustained donor engraftment at 42 days and survival at 100 days post transplantation in patients treated with anti-thymocyte globulin, clofarabine, and rituximab.

Secondary

* To determine incidence of treatment-related mortality at day 100 post transplantation.
* To determine incidence of neutrophil recovery by day 42 post transplantation.
* To determine survival at day 100 and 1 year post transplantation.
* To determine the proportion of patients with chimerism at day 28 post transplantation.
* To determine incidence and severity of grades II-IV acute graft-vs-host disease by day 100 post transplantation.

OUTLINE:

* Conditioning regimen: Patients receive rituximab intravenously (IV) on day -7, anti-thymocyte globulin IV over 4-6 hours on days -6 to -4, and clofarabine IV over 1 hour on days -4 to -2.
* Hematopoietic stem cell transplantation (HSCT): Patients undergo HSCT on day 0. Patients may receive umbilical cord blood, peripheral blood stem cells, or bone marrow from unrelated or related donors.
* Graft-vs-host disease (GVHD) prophylaxis: Patients receive oral cyclosporine twice daily or cyclosporine IV every 8 hours beginning on day -3 and continuing for 100 or 180 days post transplantation followed by a taper; mycophenolate mofetil IV every 8 hours beginning on day -3 and continuing for 30 days (or 7 days after engraftment with no evidence of GVHD); and filgrastim (G-CSF) IV once daily beginning on day 1 and continuing until blood counts recover.

After completion of study therapy, patients are followed on days 100, 180, and 360.

ELIGIBILITY:
Patient Inclusion Criteria:

* Timing of relevant evaluations: Taking in account the need for rapid intervention, if white blood count is less than 200 on day +20, bone marrow aspirate should be performed on day +21. Unless there is an increase in absolute neutrophil count (ANC) to > 500 in the following 7 days, bone marrow aspirate should be repeated on day +28. If the white blood count is still less than 200 and bone marrow is acellular, bone marrow (BM) or peripheral blood stem cell (PBSC) donor should be reactivated and availability of cord blood (CB) units assessed. If the BM or PBSC donor is not confirmed within 14 days of the request for the donation (typically second donation from the same donor), CB unit should be used instead.

Primary or secondary graft failure after hematopoietic stem cell transplantation defined as a > 50% loss of donor chimerism from previous maximum or less than 25% donor beyond day +42 with pancytopenia and no evidence of relapse. Patients with any diagnosis, type of donor, hematopoietic cell graft or conditioning regimen should be considered for this study.

* primary graft failure is defined as:

  * ANC < 500
  * BM < 10% on two occasions (Day +21 and Day +28)
  * Donor chimerism need not to be considered, provided there is no evidence of malignancy
* secondary graft failure is defined as < 5% cellularity and ANC < 500 for more than 7 days any time after primary engraftment).

  * Women of childbearing potential must agree to use adequate contraception (diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, subcutaneous implants, or abstinence, etc.) for the duration of treatment.
  * Patients or their guardian are able and willing to provide written informed consent.

Patient Exclusion Criteria:

The presence of any of the following excludes a patient from study enrollment:

* Uncontrolled active infection defined as more than one week with no response to appropriately chosen antibiotics
* Evidence of recurrence of primary malignancy.
* Pregnant or lactating. The agents used in this study may be teratogenic to a fetus and there is no information on the excretion of agents into breast milk. All females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy. Women of childbearing age must use appropriate methods as described.
* Allergy to rituximab.
* Evidence of HIV infection or positive HIV serology.
* Autologous recovery defined as defined as greater than 90% recipient PCR product in the competitive VNTR PCR performed on gradually increasing white blood cell count.

Donor Inclusion Criteria:

* Related donors must be 2-75 years of age and in good health.
* Meets match criteria
* Able and willing to undergo cell collection procedures (bone marrow cell collection or leukapheresis)
* Not pregnant or lactating.
* HIV-1, HIV-2 negative; HTLV-1, HTLV-2 negative, Hepatitis B and C negative.
* Patients or their guardian are able and willing to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-01; Primary Completion 2014-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jakub Tolar, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Conditioning for Graft Failure After Transplant: Day -7: Rituximab 375 mg/m2 Day -6: Antithymocyte globulin (Thymoglobulin) 3 mg/kg IV over 4 hours Day -5: Antithymocyte globulin (Thymoglobulin) 3 mg/kg IV over 4 hours Day -4: Clofarabine 30 mg/m2 IV over 1 hour and Antithymocyte globulin (Thymoglobulin) 3 mg/kg IV over 4 hours Day -3: Clofarabine 30 mg/m2 IV over 1 hour Day -2: Clofarabine 30 mg/m2 IV over 1 hour Day -1: Rest Day 0: Stem Cell Infusion
Period: Overall Study
Arm/Group | Conditioning for Graft Failure After Transplant
Started | 12
Completed | 11
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Conditioning for Graft Failure After Transplant
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Rate of Sustained Donor Engraftment
Description: Rate of Sustained Donor Engraftment is defined as the percent of paticipants with an absolute neutrophile count (ANC) of 500 or more without a subsequent graft rejection.
Time Frame: Day 42 post transplantation
Measure: Number; unit: percentage of participants
Arm/Group | Conditioning for Graft Failure After Transplant
Number analyzed (Participants) | 11
percentage of participants | 73

2. Primary Outcome: Survival at 100 Days Post Transplant
Description: Percent of patients alive from beginning of study to Day 100 post transplantation
Time Frame: Day 100 post transplantation
Measure: Number; unit: percentage of participants
Arm/Group | Conditioning for Graft Failure After Transplant
Number analyzed (Participants) | 11
percentage of participants | 73

3. Secondary Outcome: Treatment-related Death
Description: Percent of patients who died related to the treatment in this study.
Time Frame: Day 100 post transplantation
Measure: Number; unit: percentage of participants
Arm/Group | Conditioning for Graft Failure After Transplant
Number analyzed (Participants) | 11
percentage of participants | 18

4. Secondary Outcome: Time to Primary Neutrophil Engraftment
Description: Time to primary neutrophil engraftment is defined as the percent of patients with an absolute neutrophil count (ANC) of 500 or more neutrophils in a cubic millimeter of blood.
Time Frame: Day 42 post transplantation
Measure: Number; unit: percentage of participants
Arm/Group | Conditioning for Graft Failure After Transplant
Number analyzed (Participants) | 11
percentage of participants | 73

5. Secondary Outcome: Survival
Description: Percent of patients alive from beginning of study to one year post transplantation
Time Frame: One year post transplantation
Measure: Number; unit: percentage of participants
Arm/Group | Conditioning for Graft Failure After Transplant
Number analyzed (Participants) | 11
percentage of participants | 36

6. Secondary Outcome: Chimerism
Description: Occurrence of genetically distinct cell types in a single organism
Time Frame: Day 28 post transplantation
Measure: Median (Full Range); unit: percentage of donor cells
Arm/Group | Conditioning for Graft Failure After Transplant
Number analyzed (Participants) | 11
percentage of donor cells | 95 [0 to 100]

7. Secondary Outcome: Acute Graft-vs-host Disease
Description: Percent of patients with Acute Graft-vs-host Disease - a process where T-cells present in the donor's bone marrow at the time of transplant identify the transplant patient as "non-self' and attack the patient's skin, liver, stomach, and/or intestines.
Time Frame: Day 30-100
Measure: Number; unit: percentage of participants
Arm/Group | Conditioning for Graft Failure After Transplant
Number analyzed (Participants) | 11
percentage of participants | 18

ADVERSE EVENTS:
Arm/Group | Conditioning for Graft Failure After Transplant
Serious Adverse Events (participants affected / at risk) | 7/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Conditioning for Graft Failure After Transplant (N=11)
Graft failure (Injury, poisoning and procedural complications) | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Multi-system organ failure (General disorders) | 2
Infection (Infections and infestations) | 1
Neoplasm, malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Disease relapse
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Conditioning for Graft Failure After Transplant (N=11)
Peripheral neuropathy (Nervous system disorders) | 1
Renal failure (Renal and urinary disorders) | 5
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2
Tachycardia (Cardiac disorders) | 1
Esophageal necrosis (Gastrointestinal disorders) | 1
Gastrointestinal bleed (Gastrointestinal disorders) | 5
Cholangitis (Hepatobiliary disorders) | 1
Aseptic/avascular necrosis (Musculoskeletal and connective tissue disorders) | 1
Anxiety attacks (Psychiatric disorders) | 1
Pain NOS (General disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 8
Encephalopathy (Nervous system disorders) | 1
Osteomyelitis (Infections and infestations) | 1
Small vessel ischemia disease (Vascular disorders) | 1
Cystitis (Renal and urinary disorders) | 2
Pseudotumor cerebri (Nervous system disorders) | 1
Bradycardia (Cardiac disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Gastrointestinal infection (Infections and infestations) | 1
Bacteremia (Infections and infestations) | 2
Sepsis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Hyperdense focus in parietal lobe of brain (Nervous system disorders) | 1
Decreased brain volume (Nervous system disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Capillary leak syndrome (Vascular disorders) | 1
Partial small bowel obstruction (Gastrointestinal disorders) | 1
Viremia (Infections and infestations) | 1
Veno-occlusive disease (Vascular disorders) | 1
Hydrocephalus (Nervous system disorders) | 1
Stevens Johnson syndrome (Skin and subcutaneous tissue disorders) | 1
Vancomycin-resistant enterococci (Infections and infestations) | 1
Multi-system organ failure (Gastrointestinal disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Deep vein thrombosis vs. cellulitis (Vascular disorders) | 1
Eye hemorrhage (Eye disorders) | 1
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hemorrhagic cystitis (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes